CLINICAL TRIAL: NCT05150873
Title: Anatomical Feasibility of an Off-the-shelf Scalloped Stent-graft for Infrarenal Abdominal Aneurysm With a Hostile Neck (ReSTHoNe Study)
Brief Title: Anatomical Feasibility of an Off-the-shelf Scalloped Stent-graft for Infrarenal Abdominal Aneurysm With a Hostile Neck
Acronym: ReSTHoNe
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Responsible Party: Principal Investigator, Roberto Silingardi, MD, Associate Professor in Vascular Surgery, Chief of department, Azienda Ospedaliero-Universitaria di Modena
Other Study IDs: 3499
Record Dates: First submitted 2021-11-25; First posted 2021-12-09 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Aortic Aneurysm
Keywords: EVAR; AAA; Off-the-shelf
MeSH Terms: conditions — Aortic Aneurysm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients ttreatted for AAA: Patients affected by AAA and treated att our institution with EVAR and/or Open Repair between 2010 and 2020
  Interventions: Other: CTA evaluation

INTERVENTIONS:
Other: CTA evaluation — Any pre-operattive CTA of the patients of the cohort will be carefully evaluated to determine the theoric anatomical feasibility of an off the shelf Endograft, particularly in patients with an angulated and short aortic neck

SUMMARY:
In clinical practice a lot of EVAR cases are performed IFU for adverse neck anatomy(6) with acceptable short- and mid-term outcomes, but the long-term durability is currently an issue (7). Neck length shorter than 15 mm and angulation are two of. neck charteristics. that contribute more to define an "hostile neck" (8). The issue linked to the anatomical not feasibility of standard EVAR in patients not eligible for OR can be solved with custom made devices (CMD), but they were limited by high production costs and long time for creations (10-12 weeks)1. Nowadays no one off-the-shelf device aimed to overcome neck hostility in AAA is available on the market.

The present study aims at evaluating the anatomical applicability of an off-the-shelf scalloped stent-graft to treat infrarenal AAA with a short and/or angulated neck.

DETAILED DESCRIPTION:
Endovascular aneurysm repair (EVAR) is currently accepted as the preferred choice to treat abdominal aortic aneurysms (AAA) with feasible anatomy. Although approximately 40-60% of AAA patients are not considered anatomically feasible for EVAR, mainly in reason of a "hostile neck anatomy". In ''real-world'' clinical practice, up to 44% of EVAR cases are performed outside Instruction For Use (IFU) for adverse neck anatomy. The off-label use of standard EVAR is currently used for patients who are not eligible for OR, with acceptable short- and mid-term outcomes, Endovascular aneurysm repair (EVAR) is currently accepted as the preferred choice to treat the abdominal aortic aneurysms (AAA) with feasible anatomy. Although approximately 40-60% of AAA patients are not considered anatomically feasible for EVAR, mainly in reason of a "hostile neck anatomy"3-5. In ''real-world'' clinical practice, up to 44% of EVAR cases are performed outside Instruction For Use (IFU) for adverse neck anatomy. The off-label use of standard EVAR is currently used for patients who are not eligible for OR, with acceptable short- and mid-term outcomes, but the long-term durability of EVAR depends on the maintenance of the seal between the endograft and the aortic neck as well as the iliac arteries. Some aortic neck characteristics contribute to the definition of ''hostile neck,'' particularly length shorter than 15 mm and angulation among others. From a recent Consensus Conference, the influence of each characteristic on early or late EVAR failure is not clear, but hostile neck morphology is generally associated with higher rates of aneurysm-related adverse events and mortality. A recent independent Expert Panel, applying the Delphi methodology Indeed, agreed to define 10 mm as the threshold value below which standard EVAR should not be considered feasible. Moreover, the same experts agreed on the fact that an angulation above 60° is considered a hostile criterion for EVAR procedure. Finally should be considered that some "hostility" factors can be present at the same time and create the ideal condition for EVAR failure. The issue linked to the anatomical not the feasibility of standard EVAR in patients not eligible for OR can be solved with custom made devices (CMD), but they were limited by high production costs and long time for creations (10-12 weeks)1. Nowadays no one off-the-shelf device aimed to overcome neck hostility in AAA is available on the market.

The present study aims at evaluating the anatomical applicability of an off-the-shelf scalloped stent graft to treat infrarenal AAA with a short and/or angulated neck. From an informal review of some CTA of patients treated with EVAR or OR in mentioned unit, the authors found that more the 20% presented a distance between the two renal arteries more than 5mm. The idea of an "off-the-shelf" graft with a single scallop theoretically had to permit to gain some length along the aortic neck. Furthermore also in the case of angulation, a single scallop theoretically reduced the risk of bird beck and gutter. The aim of the study is to evaluate if a single scalloped "off-the-shelf" stent graft could be appliable and feasible in an adequate number of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients Electively treated with EVAR or AAA at the coordinator center
* Age >18
* Both sex
* Preoperative 2.5mm CTA available
* Written informed consent.

Exclusion Criteria:

* All. patients not fulfilling the inclusion criteria

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients affected by AAAs and electively treated with EVAR or OR in the Vascular Surgery Unit of Modena e Reggio Emilia from 2010 to 2020 were considered eligible for the ex-vivo feasibility study. Mandatory condittion for tthhe enrollemnt is an available 2.5mm CTA.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Anatomica feasibility and applicability of an "off-the-shelf" scallopped stent-graft measured mesured fitting three device model with data recorded from CTA of patients with AAA treted in our unit | 6-months
  observational study on the anatomical applicability in the coordinator center of an off-the-shelf scalloped device to treat infrarenal AAA with short and/or angulated neck. 3 different endograft designs were constructed. The preoperative measurements were made according to a previously described methodology. The models were matched with each preoperative CTA measure in order to evaluate if they fit or not in the index patients.

CONTACTS AND LOCATIONS:
Locations (1):
- AOU di Modena, OCB, Baggiovara, Modena, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wanhainen A, Verzini F, Van Herzeele I, Allaire E, Bown M, Cohnert T, Dick F, van Herwaarden J, Karkos C, Koelemay M, Kolbel T, Loftus I, Mani K, Melissano G, Powell J, Szeberin Z, Esvs Guidelines Committee, de Borst GJ, Chakfe N, Debus S, Hinchliffe R, Kakkos S, Koncar I, Kolh P, Lindholt JS, de Vega M, Vermassen F, Document Reviewers, Bjorck M, Cheng S, Dalman R, Davidovic L, Donas K, Earnshaw J, Eckstein HH, Golledge J, Haulon S, Mastracci T, Naylor R, Ricco JB, Verhagen H. Editor's Choice - European Society for Vascular Surgery (ESVS) 2019 Clinical Practice Guidelines on the Management of Abdominal Aorto-iliac Artery Aneurysms. Eur J Vasc Endovasc Surg. 2019 Jan;57(1):8-93. doi: 10.1016/j.ejvs.2018.09.020. Epub 2018 Dec 5. No abstract available. PMID 30528142
- [Background] Gimenez-Gaibar A, Gonzalez-Canas E, Solanich-Valldaura T, Herranz-Pinilla C, Rioja-Artal S, Ferraz-Huguet E. Could Preoperative Neck Anatomy Influence Follow-up of EVAR? Ann Vasc Surg. 2017 Aug;43:127-133. doi: 10.1016/j.avsg.2016.12.011. Epub 2017 Apr 6. PMID 28390913
- [Background] Caradu C, Berard X, Midy D, Ducasse E. Influence of Anatomic Angulations in Chimney and Fenestrated Endovascular Aneurysm Repair. Ann Vasc Surg. 2017 Aug;43:104-114. doi: 10.1016/j.avsg.2017.01.002. Epub 2017 Feb 28. PMID 28258015
- [Background] Speziale F, Sirignano P, Setacci F, Menna D, Capoccia L, Mansour W, Galzerano G, Setacci C. Immediate and two-year outcomes after EVAR in "on-label" and "off-label" neck anatomies using different commercially available devices. analysis of the experience of two Italian vascular centers. Ann Vasc Surg. 2014 Nov;28(8):1892-900. doi: 10.1016/j.avsg.2014.06.057. Epub 2014 Jul 7. PMID 25011083
- [Background] Muhs BE, Jordan W, Ouriel K, Rajaee S, de Vries JP. Matched cohort comparison of endovascular abdominal aortic aneurysm repair with and without EndoAnchors. J Vasc Surg. 2018 Jun;67(6):1699-1707. doi: 10.1016/j.jvs.2017.10.059. Epub 2017 Dec 18. PMID 29248241
- [Background] AbuRahma AF, DerDerian T, AbuRahma ZT, Hass SM, Yacoub M, Dean LS, Abu-Halimah S, Mousa AY. Comparative study of clinical outcome of endovascular aortic aneurysms repair in large diameter aortic necks (>31 mm) versus smaller necks. J Vasc Surg. 2018 Nov;68(5):1345-1353.e1. doi: 10.1016/j.jvs.2018.02.037. Epub 2018 May 22. PMID 29802043
- [Background] Chaikof EL, Fillinger MF, Matsumura JS, Rutherford RB, White GH, Blankensteijn JD, Bernhard VM, Harris PL, Kent KC, May J, Veith FJ, Zarins CK. Identifying and grading factors that modify the outcome of endovascular aortic aneurysm repair. J Vasc Surg. 2002 May;35(5):1061-6. doi: 10.1067/mva.2002.123991. No abstract available. PMID 12021728
- [Background] Marone EM, Freyrie A, Ruotolo C, Michelagnoli S, Antonello M, Speziale F, Veroux P, Gargiulo M, Gaggiano A. Expert Opinion on Hostile Neck Definition in Endovascular Treatment of Abdominal Aortic Aneurysms (a Delphi Consensus). Ann Vasc Surg. 2020 Jan;62:173-182. doi: 10.1016/j.avsg.2019.05.049. Epub 2019 Aug 6. PMID 31394211
- [Background] Gallitto E, Faggioli G, Spath P, Pini R, Mascoli C, Ancetti S, Stella A, Abualhin M, Gargiulo M. The risk of aneurysm rupture and target visceral vessel occlusion during the lead period of custom-made fenestrated/branched endograft. J Vasc Surg. 2020 Jul;72(1):16-24. doi: 10.1016/j.jvs.2019.08.273. Epub 2020 Feb 13. PMID 32063442
- [Result] Chaikof EL, Dalman RL, Eskandari MK, Jackson BM, Lee WA, Mansour MA, Mastracci TM, Mell M, Murad MH, Nguyen LL, Oderich GS, Patel MS, Schermerhorn ML, Starnes BW. The Society for Vascular Surgery practice guidelines on the care of patients with an abdominal aortic aneurysm. J Vasc Surg. 2018 Jan;67(1):2-77.e2. doi: 10.1016/j.jvs.2017.10.044. PMID 29268916

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/73/NCT05150873/Prot_SAP_000.pdf